CLINICAL TRIAL: NCT02878889
Title: A Phase II Trial of S-1 as Maintenance Treatment After Gemcitabine Plus Cisplatin Regimen Chemotherapy in Patients With Recurrent and/or Metastatic Nasopharyngeal Carcinoma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-16-01
Record Dates: First submitted 2016-08-15; First posted 2016-08-25 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — S 1 (combination)

ARMS (1):
- Arm 1 (Experimental): S-1 as Maintenance Treatment After Gemcitabine Plus Cisplatin Regimen Chemotherapy in Patients With Recurrent and/or Metastatic Nasopharyngeal Carcinoma.
  Interventions: Drug: S-1

INTERVENTIONS:
Drug: S-1

SUMMARY:
A Phase II Trial of S-1 as Maintenance Treatment After Gemcitabine Plus Cisplatin Regimen Chemotherapy in Patients With Recurrent and/or Metastatic Nasopharyngeal Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* all proven to have locoregional recurrence after curative treatment and unsuitability for further local treatment, distant metastases at presentation or acquired metastases after curative treatment. the presence of at least one measurable disease, which was defined as lesion that could be measured at least 20 mm in one dimension by conventional computed tomography (CT) or at least 10 mm by spiral CT scan; KPS≥70, and a life expectancy of at least 6 months.

Exclusion Criteria:

* other malignancy prior to study entry; bone-only metastasis;previous radiotherapy within 4 weeks; previous exposure to gemcitabine;patients with any active, non-controlled infection or other severe systemic diseases, such as congestive heart failure, angina pectoris, respiratory insufficiency and arrhythmia were all rejected at enrollment. Other exclusion criteria included concurrent treatment with other investigational drugs, hypersensitivity to platinum compounds,and current pregnancy or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xiaozhong Chen, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang